CLINICAL TRIAL: NCT04433377
Title: Comparison of the Effects of Ultrasound-guided Suprascapular Nerve Block and Subacromial Injection in Hemiplegic Shoulder Pain: a Randomized Controlled Trial
Brief Title: Comparison Suprascapular Nerve Block and Subacromial Injection in Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Corum, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-118
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Hemiplegia; Pain
MeSH Terms: conditions — Hemiplegia; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprascapular nerve block group (Experimental): Suprascapular nerve block will be performed with a MyLab60 model a high resolution 7-12-MHz linear probe ultrasonography device. After the suprascapular fossa will be observed by ultrasonography, a betamethasone dipropionate plus betamethasone sodium phosphate solution (6.43 mg / mL + 2.63 mg / mL; 1 mL), 0.5 % bupivacaine (2 mL) and physiological serum (2 mL) will be injected with an in-plane technique using a 22 gauge 90-mm injector.
  Home exercise: The exercise program consists of passive and active-assistive ROM exercises (3 sets daily, 20 times in each set).
  Interventions: Procedure: Suprascapular nerve block
- Subacromial injection group (Experimental): Subacromial injection will be performed with a MyLab60 model a high resolution 7-12-MHz linear probe ultrasonography device. After the subacromial bursa will be observed by ultrasonography, a betamethasone dipropionate plus betamethasone sodium phosphate solution (6.43 mg/mL + 2.63 mg/mL; 1 mL), 2% lidocaine (2 mL) and physiological serum (2 mL) will be injected with an in-plane technique using a 21 gauge 38-mm injector.
  Home exercise: The exercise program consists of passive and active-assistive ROM exercises (3 sets daily, 20 times in each set).
  Interventions: Procedure: Subacromial injection

INTERVENTIONS:
Procedure: Suprascapular nerve block — A betamethasone dipropionate plus betamethasone sodium phosphate solution (6.43 mg / mL + 2.63 mg / mL; 1 mL), 0.5 % bupivacaine (2 mL) and physiological serum (2 mL) are injected with an in-plane technique using a 22 gauge 90-mm injector
  Arms: Suprascapular nerve block group
Procedure: Subacromial injection — A betamethasone dipropionate plus betamethasone sodium phosphate solution (6.43 mg/mL + 2.63 mg/mL; 1 mL), 2% lidocaine (2 mL) and physiological serum (2 mL) are injected with an in-plane technique using a 21 gauge 38-mm injector.
  Arms: Subacromial injection group

SUMMARY:
Hemiplegic shoulder pain is the most common poststroke painful condition. Hemiplegic shoulder pain reduces range of motion (ROM) and hand function, resulting in limited daily life activity and decreased quality of life.

In the literature, the effectiveness of suprascapular nerve block and subacromial injection in hemiplegia patients with shoulder pain has been previously evaluated, but these injection treatments have not been compared.

Therefore, the aim of this study is to compare the effectiveness of suprascapular nerve block and subacromial injection on pain, shoulder (ROM), function and quality of life in hemiplegia patients with shoulder pain.

DETAILED DESCRIPTION:
Patients will be randomly assigned Subacromial injection group or Suprascapular nerve block group

In the suprascapular nerve block group, suprascapular nerve block will be performed with a MyLab60 model a high resolution 7-12-MHz linear probe ultrasonography device. After the suprascapular fossa will be observed by ultrasonography, a betamethasone dipropionate plus betamethasone sodium phosphate solution (6.43 mg / mL + 2.63 mg / mL; 1 mL), 0.5 % bupivacaine (2 mL) and physiological serum (2 mL) will be injected with an in-plane technique using a 22 gauge 90-mm injector.

In the subacromial injection group, subacromial injection will be performed with a MyLab60 model a high resolution 7-12-MHz linear probe ultrasonography device. After the subacromial bursa will be observed by ultrasonography, a betamethasone dipropionate plus betamethasone sodium phosphate solution (6.43 mg/mL + 2.63 mg/mL; 1 mL), 2% lidocaine (2 mL) and physiological serum (2 mL) will be injected with an in-plane technique using a 21 gauge 38-mm injector.

A home exercise program will be given both groups. The exercise program consisted of passive and active-assistive ROM exercises (3 sets daily, 20 times in each set).

ELIGIBILITY:
Inclusion Criteria:

* Brunstrom stage 2 to 5
* spasticity <4 according to the modified Ashworth scale
* having hemiplegia less than 12 months
* Presence of shoulder pain lasting more than 3 months
* Conservative treatment for painful shoulder before injection

Exclusion Criteria:

* Patients over 75 years old, under 30 years old
* Anti-coagulant or antiaggregant use
* Presence of diabetes mellitus
* Patients who could not be cooperated and Mini-mental Test (MMSE) score <24
* Having previously had suprascapular block or subacromial injection
* Presence of complex regional pain syndrome (type I),
* The presence of neglect syndrome

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Visual Analog Scale (VAS) score | baseline, month 1 and month 3
  Self-reported neck pain intensity will be evaluated with the Visual Analog Scale (VAS). Patients will be asked about the average pain intensity that they had felt in the past week ("0" defines "no pain" and "10" defines "unbearable pain'').

SECONDARY OUTCOMES:
Shoulder ROM | baseline, month 1 and month 3
  The shoulder ROM (flexion, abduction, internal rotation, external rotation) will be passively assessed by goniometry.
Functional Independence Measure (FIM) | baseline, month 1 and month 3
  Functional independence measure (FIM) will be used to evaluate independence for the activities of daily living. It was developed to measure the results of the rehabilitation on the patient. The higher scores in FIM are interpreted as better functional independence
EuroQol 5D-3L questionnaire (EQ-5D-3L) | baseline, month 1 and month 3
  The EQ-5D-3L scale, which scores five health conditions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) through evaluation at 3 levels (no problems, some problems, or extreme problems), will be used to evaluate the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Corum, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No